CLINICAL TRIAL: NCT03123458
Title: Clonal Fetal Mesenchymal Stem Cells (cfMSCs) for the Control of Immune-related Disorders
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Responsible Party: Principal Investigator, Lung-Ji Chang, President, Shenzhen Geno-Immune Medical Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-17001
Record Dates: First submitted 2017-03-13; First posted 2017-04-21 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-09

CONDITIONS: Immune Related Disorder; Tissue Damage
Keywords: MSC; GVHDs; transplantation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm, cfMSC to treat immune disorders (Experimental): cfMSCs treatment
  Interventions: Biological: clonal fetal MSCs

INTERVENTIONS:
Biological: clonal fetal MSCs — clonal fetal MSCs

SUMMARY:
The primary objectives are to evaluate the safety and efficacy of infusion of the third party fully-characterized clonally derived fetal MSCs (cfMSCs) for the control of severe symptoms associated with acute and chronic immune-related disorders and tissue damage.

DETAILED DESCRIPTION:
MSCs have been extensively studied and clinically evaluated for the treatment of autoimmune diseases and graft versus host disease (GVHD) after hematopoietic stem cell transplantation (HSCT). The variable source of MSCs and the lack of consistency of primary tissue-derived MSCs are major obstacles to reliable translational applications of such therapeutic cell products. Fetal tissue-derived clonal MSCs (cfMSCs) have extended expansion potential and express rich levels of various growth factors, and thus can achieve quality consistency. Careful evaluation of fMSCs in clinical studies has not been conducted. Autoimmune diseases involve aberrant immune responses that harm tissues and organs. GVHD is a serious and often fatal problem associated with HSCT. MSCs have immunomodulatory and immunosuppressive effects. In many studies, MSCs have demonstrated promising beneficial effects that reduce severe autoimmune reactions, diminish symptoms of chronic GvHD and therapy-resistant acute GvHD including steroid-resistant GVHD. The safety and therapeutic effects of phenotype and functionally characterized fMSCs still require extensive clinical evaluation. This study aims to assess the safety and the potential beneficial effects of infusion of various dosages of third party fMSCs for the control of severe symptoms associated with acute and chronic immune-related disorders.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent.
2. No available alternative treatment that can reduce the symptoms
3. Patients are required to meet the following inclusion criteria:

   * Any patient that has clinically documented abnormal immune or age-related disorders including acute and chronic GVHD. Patients may receive best available treatment for the control of disease symptoms.
   * Patients with symptoms associated with genetic defects or infectious diseases are not eligible.

Exclusion Criteria:

1. Inability to give informed consent.
2. Patients with ongoing infection or history of cancer.
3. Patients with poor clinical conditions with the life expectancy of less than 14 days.
4. Pregnancy.

Ages: 1 Year to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | up to one month
  Safety of cfMSC infusion acute and prolonged

SECONDARY OUTCOMES:
Number of participants with reduced symptoms or stabilized conditions after treatment | after 1 month from fMSC infusion
  Short term clinical effects measured by physiological and serological parameters related to the disease condition and symptoms using prepared study assessment table.

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Capital Institute of Pediatrics affiliated Children's hospital, Beijing, Beijing Municipality
  - Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong
  - Aerospace Center Hospital, Beijing